CLINICAL TRIAL: NCT05332678
Title: An Open-Label, Proof-of-Concept Study to Evaluate the Safety and Treatment Effects of SLS-005 (Trehalose Injection, 90.5 mg/mL for Intravenous Infusion) in Participants With Alzheimer's Disease (AD)
Brief Title: SLS-005 (Trehalose Injection) in the Treatment of Alzheimer's Disease
Acronym: [STRIVE-AD]
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Seelos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLS-005-207
Record Dates: First submitted 2022-03-25; First posted 2022-04-18 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer's Disease
Keywords: Trehalose; Phase II; Dementia; Australia; SLS-005; STRIVE-AD
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLS-005 - Once Weekly (Experimental): SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion). SLS-005 will be administered as a weight-based dose of 0.75 g/kg by IV infusion once a week over 60 ± 5 minutes for volumes <600 mL or 90 minutes +5 min for volumes >600 mL.
  For 52 weeks.
  Interventions: Drug: SLS-005 - Once Weekly
- SLS-005 - Twice Weekly (Experimental): SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion). SLS-005 will be administered as a weight-based dose of 0.75 g/kg by IV infusion twice a week over 60 ± 5 minutes for volumes <600 mL or 90 minutes +5 min for volumes >600 mL.
  For 52 weeks.
  Interventions: Drug: SLS-005 - Twice Weekly

INTERVENTIONS:
Drug: SLS-005 - Once Weekly — Please see Arm description.
  Other Names: SLS-005
  Arms: SLS-005 - Once Weekly
Drug: SLS-005 - Twice Weekly — Please see Arm description.
  Other Names: SLS-005
  Arms: SLS-005 - Twice Weekly

SUMMARY:
An open-label, proof-of-concept study to evaluate the safety and treatment effects of SLS-005 in Participants with Alzheimer's Disease (AD) treated once or twice weekly for 52 weeks.

DETAILED DESCRIPTION:
This is an open-label proof-of-concept study to evaluate the safety and treatment effects of SLS-005 (trehalose injection, 90.5 mg/mL for intravenous infusion) administered by IV infusion in either a once weekly or twice weekly dosing regimen in eligible men and women, ages 50-85 years, who have very mild, mild, or moderate dementia as determined by the Clinical Dementia Rating (CDR) global score and a biomarker-supported diagnosis of AD guided by the National Institute on Aging and Alzheimer's Association (NIA-AA) Research Framework.

The study will enroll approximately 30 eligible participants who will be assigned in a 1:1 ratio to treatment with SLS-005 at a dose of 0.75 g/kg. administered by intravenous (IV) infusion in either a once weekly or twice weekly dosing regimen for up to 52 weeks. Participants will be assigned to 1 of the 2 dosing regimens to achieve approximately equal numbers of participants with mild (CDR 0.5 or 1) and moderate (CDR 2) baseline dementia severity in each dosing regimen. A relatively equal number of participants enrolled in each dosing regimen will be assigned to either the amyloid or tau PET procedure. Tracers to be used will be approved by Sponsor and described in the imaging manual.

Adverse events and results of laboratory and physical evaluations will be collected and assessed throughout the study. Fluid biomarkers associated with AD pathology, brain imaging including amyloid or tau PET and volumetric magnetic resonance imaging (MRI), and measures of cognitive performance, functioning in activities of daily living (ADL), and neuropsychiatric behavioral symptoms will be collected at baseline and at scheduled times throughout the study. Participants who terminate treatment early, will be encouraged to complete all safety and outcome procedures as specified in the protocol's schedule of events.

ELIGIBILITY:
Inclusion Criteria

1. Have a study partner/caregiver who, in the Investigator's judgment, has frequent and sufficient face-to-face contact with the participant (approximately 10 hours per week or more) and consents to attend all study visits, assist in ensuring compliance with all study requirements and procedures, and provide input into assessments of cognitive performance and functioning in daily activities throughout the full duration of the participant's involvement in the study.
2. Signed informed consent from:

   1. The participant or person responsible/guardian
   2. The participant's study partner/caregiver
3. Men and women, 50 to 85 years (inclusive) of age.
4. Gradual and progressive change in cognitive performance has been observed for ≥ 6 months not associated with a specific event or medical condition e.g., head trauma, stroke, cardiac arrest, cerebrovascular disease, epilepsy, alcohol abuse, etc.
5. Capable of completing study assessments either alone or with assistance from the study partner.
6. Mini-mental status examination (MMSE) score ≥ 16 and ≤ 27 at screening.
7. Modified Hachinski Score ≤ 4 at screening.
8. Body Mass Index (BMI) between 20 kg/m2 and 32 kg/m2 (inclusive)
9. Clinical Dementia Rating (CDR) global score of 0.5, 1.0, or 2.0 at screening.
10. Clinical Dementia Rating - Sum of Boxes (CDR-SB) score ≥ 0.5 at screening.
11. Documentation of results for either CSF Aβ42, CSF Aβ42/Aβ40 ratio, or brain imaging with PET (amyloid or tau) that was consistent with a diagnosis of AD within 12 months of screening.
12. Stable doses of all concomitant medications for at least 30 days prior to the baseline visit.
13. For participants taking cholinesterase inhibitors and/or memantine, documentation of stable use for at least 12 weeks is required prior to screening.
14. Negative serum beta-human chorionic gonadotropin (ß-hCG) pregnancy result at the screening visit for female participants of childbearing potential.
15. Willingness to comply with sexual abstinence or contraception guidelines of this study.
16. Willingness and ability to complete all study procedures, including brain magnetic resonance imaging (MRI), lumbar puncture, clinical genotyping, and brain positron emission tomography (PET).
17. Participant and study partner/caregiver must be fluent in the English language for both reading and speaking.
18. Participant and study partner/caregiver must be fully vaccinated as per local regulations for COVID-19 at least 2 weeks prior to screening.

Exclusion Criteria

1. Presence of a neurologic or neuropsychiatric condition or imaging finding associated with a neurologic or neuropsychiatric condition other than AD that can be associated with dementia or confound the evaluation of dementia, including but not limited to Parkinson's disease, Huntington's disease, frontotemporal dementia, cerebrovascular disease, (diseases related to or events associated with disruption of blood flow to the brain), seizure disorders, inflammatory or infectious disorders of the central nervous system, normal pressure hydrocephalus, traumatic brain injury, uncontrolled major depression, psychosis, bipolar disorder, and long-term sequelae of alcohol or substance abuse.
2. History of stroke or transient ischemic attack (TIA) within 12 months of screening.
3. Epileptic or epileptiform seizure within 12 months of screening.
4. Current participation in another clinical trial or completed participation in an interventional trial less than 30 days prior to the screening visit (90 days for a biological treatment).
5. Involvement in an Aβ or tau vaccination trial for AD unless known to have received only placebo.
6. Current diagnosis and/or healthcare professional-recommended treatment (medication and/or diet) of diabetes mellitus type 1 or type 2.
7. Hemoglobin A1c (HbA1c) ≥ 6.5% at the screening visit
8. Prior treatment with SLS-005, any other IV trehalose formulation, or known hypersensitivity to trehalose.
9. Is receiving aducanumab or any other immunotherapy for treatment of dementia including AD.
10. Regular use (≥ 3 days per week) of prescribed or pharmacy-purchased opiates, opioids, or benzodiazepines.
11. Pregnant or breastfeeding.
12. History of alcohol or drug abuse within the last 2 years.
13. Chronic liver disease including Hepatitis B; Hepatitis C unless successful curative treatment is documented; human immunodeficiency virus (HIV) infection.
14. Prior history of drug-induced liver injury (DILI) and/or laboratory results at screening that indicate inadequate liver function (e.g., alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase [GGT] > 2 times the upper limit of normal [x ULN] and/or total bilirubin level > 2 x ULN).
15. Laboratory results at screening that indicate inadequate renal function (e.g., estimated creatinine clearance of < 60 mL/min calculated by the Cockcroft and Gault formula).
16. Recent history of heart failure or unexplained edema or any current cardiovascular disease or abnormality on 12-lead ECG at screening that, in the investigator's opinion, is clinically significant and could be a potential safety risk to the participant, including risk factors for stroke (e.g., atrial fibrillation, cardiomyopathy).
17. History of cancer (currently active or in remission) within 5 years prior to screening, excluding treated basal or squamous skin cancer, or stable prostate cancer.
18. Lack of reliable venous access for the weekly administration of study drug.
19. Contraindications to the lumbar puncture (LP) procedure such as prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelet count < 100,000, use of an anticoagulant (e.g., warfarin), or history of a bleeding disorder.
20. Any current psychiatric or neurological disorder other than AD that, in the investigator's opinion, may interfere with the participant's ability to provide informed consent or appropriately complete the study's safety or efficacy assessments.
21. Significant suicide risk as indicated by a "yes" response to #4 or #5 under Suicidal Ideation or any "yes" response under Suicidal Behavior on the Columbia Suicide Severity Rating Scale (C-SSRS) during the screening visit.
22. Any other medical condition or abnormal finding during screening that, in the investigator's opinion, could confound collection or interpretation of safety or efficacy data or be a potential safety risk to the participant.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Endpoints for Safety and Tolerability of Treatment | over 52 week treatment period
  Incidences of treatment-emergent Adverse Events and Serious Adverse Events (SAEs), including clinically significant laboratory and electrocardiogram (ECG) abnormalities
Endpoints for Safety and Tolerability of Treatment | 52 weeks
  Incidences of treatment-emergent early study and treatment discontinuations.

SECONDARY OUTCOMES:
Endpoints for Treatment Effects on Imaging Biomarkers Associated with AD | 26 and 52 weeks
  Changes in brain imaging biomarkers associated with AD
Endpoints for Treatment Effects on CSF Biomarkers Associated with AD | 26 and 52 weeks
  Changes in CSF biomarkers associated with AD
Endpoints for Treatment Effects on Volumes of Brain Structures | 26 and 52 weeks
  Changes in the volumes of specified brain structures as measured by brain MRI
Exploratory Endpoints - Treatment Effects in Cognitive Performance | 13, 26, 39 and 52 weeks
  Changes from baseline in cognitive performance as measured by the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog 13). ADAS-Cog 13 is a series of questions to the participant and tasks for the participant to perform. It is used to measure cognitive functions and non-cognitive functions such as mood and behaviour
Exploratory Endpoints - Treatment Effects in Dementia Severity | 13, 26, 39 and 52 weeks
  Changes from baseline in dementia severity as measured by the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB). The CDR-SB is a semi structured interview with the participants caregiver, used to asses the severity of the symptoms of dementia.
Exploratory Endpoints - Treatment Effects in Activities of Daily Living | 13, 26, 39 and 52 weeks
  Changes from baseline in functioning in activities of daily living (ADL) as measured by the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living (ADCS-iADL). The scale is used to assess functional decline in participants. The participants study partner is asked questions about the participants activities of daily living.
Exploratory Endpoints - Treatment Effects in Behavioral Symptoms and Functioning | 13, 26, 39 and 52 weeks
  Changes from baseline in behavioral symptoms and functioning as measured by the Neuropsychiatric Inventory (NPI). The purpose of the NPI is to obtain information on the presence of psychopathology in patients with brain disorders.The participants caregiver is asked questions in an interview to evaluate the participants behaviour.
Exploratory Endpoints - Treatment Effects in Cognitive Impairment | 26 and 52 Weeks.
  Change from baseline in Mini-mental status examination (MMSE). The rater will ask the participant a series of questions and ask the participants to perform some tasks. It used to assess cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Neurodegenerative Disorders Research Pty Ltd, West Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No